CLINICAL TRIAL: NCT01985178
Title: Omega-3 Fatty Acids as Adjunctive Treatment for Adolescents With Eating Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12345
Record Dates: First submitted 2013-09-19; First posted 2013-11-15 (Estimated); Last update posted 2020-12-22 (Actual); Status verified 2015-04

CONDITIONS: Eating Disorder
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Omega-3 Fatty Acid Supplement (Experimental)
  Interventions: Dietary Supplement: Omega-3 Fatty Acid Supplement

INTERVENTIONS:
Dietary Supplement: Omega-3 Fatty Acid Supplement

SUMMARY:
Eating disorders are conditions that are defined by abnormal eating habits that involve insufficient or excessive food intake. With regards to treating these disorders, there is an increasing interest in fat deprivation due to a lack of proper diet, particularly dietary fats such as polyunsaturated fatty acids. These fatty acids are essential components of the brain and are important for normal functioning of the body. Since the body cannot synthesize these fats, it has to rely completely on diet to obtain a sufficient amount. Hence, diets that lack sufficient fats or under fasting conditions, the imbalance of these fats can severely alter brain functions. The investigators want to see if these supplements are well tolerated and accepted by adolescent patients with eating disorders.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Eating Disorder, less than 18 years of age

Exclusion Criteria:

* unable to read and understand English

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2013-10; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Dropout rate | 2 months

SECONDARY OUTCOMES:
Rate of patients reporting side effects | 2 months
Change in weight | 2 months

OTHER OUTCOMES:
Severity of depressive symptoms | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Couturier, MD, Principal Investigator — McMaster University
Locations (1):
- McMaster Children's Hospital, Hamilton, Ontario, Canada